CLINICAL TRIAL: NCT02523547
Title: PhaseIVstudy to Evaluate the Non-inferiority of Cavir®Tab. in Terms of Hepatitis B Virus(HBV)DNA Undetectability Comparing Baraclude® Tab. in Hepatitis B e Antigen(HBeAg)(+) Chronic Hepatitis B Patients Treated With Long-term Baraclude® Tab
Brief Title: Study to Evaluate the Non-inferiority of Cavir in HBeAg(+)Chronic Hepatitis B Patients Treated With Baraclude
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-CAV-401
Record Dates: First submitted 2015-07-26; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Hepatitis B
Keywords: entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cavir (Experimental): entecavir/0.5mg/day
  Interventions: Drug: Cavir
- Baraclude (Active Comparator): entecavir/0.5mg/day
  Interventions: Drug: Baraclude

INTERVENTIONS:
Drug: Cavir — 0.5mg/day
  Other Names: entecavir
  Arms: Cavir
Drug: Baraclude — 0.5mg/day
  Other Names: entecavir
  Arms: Baraclude

SUMMARY:
Open-labeled, Prospective, Randomized, Multi-center, Interventional, Phase IV study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the non-inferiority and safety in terms of HBV DNA undetectability comparing Baraclude Tab. in HBeAg(+) chronic hepatitis B patients treated with long-term Baraclude Tab.

ELIGIBILITY:
Inclusion Criteria:

* Patients (over the19 years of age) currently taking Baraclude® monotherapy for chronic HBV infection for at least 24 month with < HBV DNA 60 IU/mL level, HBeAg positive and HBeAb negative status at screening.

Exclusion Criteria:

* Patients are diagnosed Hepatitis cancer and hepatocellular carcinoma (HCC)
* Patient has concomitant other chronic viral infection (HAV/Hepatitis C Virus (HCV)/Hepatitis D Virus(HDV)/HIV)
* Patient had documented resistance mutations at any time before or at screening
* Patient has clinically confirmed alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency and Wilson's Disease.
* Patient has received antiviral agent including interferon other than Baraclude within 24 months before screening for this study.
* Patient has received immunosuppressive agent within 24 weeks before screening or corticosteroids for 4 weeks.
* Clinical signs as indicated by any one of the following: Ccr(Cockroft-Gault) < 50ml/min, Total bilirubin > 3.0 mg/dl, Albumin < 2.7 g/dl, Prothrombin time > INR 2.3
* Patient is pregnant or breastfeeding or willing to be pregnant
* Patient has malignancy except for thyroid cancer and Borderline malignancy.a history of treated malignancy is allowable if the patient's malignancy has been in complete remission, off chemotherapy and without additional surgical intervention, during the preceding five years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with maintenance of HBV DNA undetectability | 48weeks
  analysis

SECONDARY OUTCOMES:
The proportion of patients with HBeAg seroconversion | at week 12, 24, 36 and 48 of treatment
  analysis
The proportion of patients with HBeAg seroclearance | at week 12, 24, 36 and 48 of treatment
  analysis
The proportion with HBsAg seroclearance | at week 48 of treatment
  analysis
The proportion with HBeAg seroconversion and HBsAb positive | at week 48 of treatment
  analysis
Changes in serum HBV DNA levels | at week 48 of treatment
  analysis
Changes in HBsAg titer | at week 48 of treatment
  analysis
Changes in ALanine amino Transferase (ALT) | at week 48 of treatment
  analysis
Proportion of patients with virologic breakthrough | at week 48 of treatment
  virologic breakthrough is defined as the increase in serum HBV DNA (>60IU/ml) as determined by at least 2 consecutive measurements of at least 3 month apart, during continued treatment
Changes in EuroQoL Five Dimensions Questionnaire-3L(EQ-5D-3L) | at week 48 of treatment
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- 15 Sites, Seoul, South Korea